CLINICAL TRIAL: NCT02001974
Title: Phase Ib Pilot Study to Evaluate Reparixin in Combination With Chemotherapy With Weekly Paclitaxel in Patients With HER 2 Negative Metastatic Breast Cancer (MBC)
Brief Title: Pilot Study to Evaluate Reparixin With Weekly Paclitaxel in Patients With HER 2 Negative Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP0111
Record Dates: First submitted 2013-11-15; First posted 2013-12-05 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Breast Cancer
Keywords: HER 2 negative; metastatic breast cancer; Cancer Stem Cells
MeSH Terms: conditions — Breast Neoplasms | interventions — Chromosomes, Artificial, P1 Bacteriophage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15 of 28-day cycle) + reparixin oral 400 mg three times daily (t.i.d.) three weeks on one week off (three to six patients)
  Interventions: Drug: Paclitaxel+Reparixin
- Group 2 (Experimental): Paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15 of 28-day cycle) + reparixin oral 100% increase to 800 mg t.i.d. if no toxicity in previous group (400 mg) three weeks on one week off (three to six patients)
  Interventions: Drug: Paclitaxel+Reparixin
- Group 3 (Experimental): Paclitaxel 80 mg/m2 i.v. (Days 1, 8, and 15 of 28-day cycle) + reparixin oral 50% increase to 1200 mg t.i.d. if no toxicity in previous group (800 mg) three weeks on one week off (three to six patients).
  Interventions: Drug: Paclitaxel+Reparixin

INTERVENTIONS:
Drug: Paclitaxel+Reparixin — Association of Paclitaxel at fixed dosage with three increasing dosage of Reparixin
  Other Names: PAC + REP

SUMMARY:
This is a phase I study to evaluate the safety and define the pharmacokinetic (PK) profile of orally administered reparixin in combination with paclitaxel in HER 2 (Human epidermal growth factor receptor-2) negative metastatic breast cancer patients.

The primary objective of this study was to evaluate the safety and define the pharmacokinetic (PK) profile of orally administered reparixin in combination with paclitaxel in HER-2 negative MBC patients.

The secondary objectives were to:

1. Evaluate the effects of orally administered reparixin on cancer stem cell (CSC) markers, the tumoral microenvironment and markers of cytokine inflammation;
2. Evaluate peripheral blood samples for enumeration of circulating tumor cells (CTCs), molecular characterization as CSCs and perform epithelial-mesenchymal transition (EMT) biomarker profiling;
3. Assess disease response for indication of efficacy.

DETAILED DESCRIPTION:
The CSC (Cancer stem cell) concept has important implications for understanding carcinogenesis as well as for the development of cancer therapeutics. According to this concept, tumors are initiated and maintained by a cellular subcomponent that displays stem cell properties. These properties include self-renewal, which drives tumorigenesis, and differentiation (albeit aberrant), which contributes to tumor cellular heterogeneity. The existence of CSCs has been described in a variety of hematologic and solid tumors including those of the breast, brain, colon, pancreas, lung, liver, and head and neck. In addition to driving tumorigenesis, CSCs may contribute to tumor metastasis as well as to tumor recurrence after treatment.

One of the therapeutic strategies being pursued to target CSCs involves inhibition of self renewal or survival pathways in these cells. These pathways include NOTCH (Notch signaling pathway), Hedgehog, and WNT (Wnt signaling pathway). Such strategies may be limited by the role of these pathways in normal stem cell function, which could result in systemic toxicities from pathway inhibition. In addition to intrinsic pathways regulating stem cell functions, normal and malignant stem cells are regulated by extrinsic signals generated in the microenvironment or CSC niche. In the breast, this niche is composed of immune cells, mesenchymal elements that include fibroblasts, endothelial cells, adipocytes, and extracellular matrix components. These components play an important role in normal breast development and carcinogenesis. If the cellular microenvironment plays an important role in the regulation of CSC growth and survival, then strategies aimed at interfering with these interactions represent a rational approach to target breast CSCs.

There are limited data on the impact of treatment tailoring based on CSCs detection. Gene profiling of CSCs could lead to identification of therapeutic targets on CSCs (e.g. hormone receptors, HER-2 [Human epidermal growth factor receptor-2] expression, EGFR [Epidermal growth factor receptor] expression), and could represent tumor biopsy in "real time". Several groups showed frequent discordance of HER-2 status between primary tumor and CSCs, and case reports showed clinical utility to use of trastuzumab-based therapy based on HER-2 CSCs status. Similarly, the hormonal status of CSCs could be different from that of the primary tumor, which could lead to increase the number of patients suitable for endocrine therapy, but also could explain why endocrine therapy fails in a subset of hormone receptor-positive patients. The study provided the in vivo demonstration that CXCR-1 (Chemokine receptor 1) targeting with specific blocking antibodies or reparixin is associated with reduced systemic metastases. The experimental data provides another therapeutic target in metastatic disease and warrants a pilot study investigation in humans to further explore effects of reparixin on breast CSCs and the tumoral microenvironment.

Reparixin seems to be a good candidate for use in breast cancer patients because of its very acceptable toxicity profile shown in the Phase I and II clinical trials conducted so far, along with its observed activity in vitro against breast cancer cell lines and in vivo in tumor xenografts in mice. It potentially addresses another therapeutic target in metastatic disease. The current pilot study thus aims at exploring the safety and PK profile of orally administered reparixin in HER-2 negative metastatic breast cancer patients and its effects on breast CSC markers.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 years.
2. Patients with histologic or cytologic diagnosis of breast cancer with evidence of metastatic disease with documented HER-2 negative status and eligible for treatment with paclitaxel.
3. Patients with at least one baseline measurable lesion according to RECIST version 1.1 criteria.
4. Zubrod (Eastern Co-operative Oncology Group [ECOG]) Performance Status (PS) of 0-1.
5. An electrocardiogram (ECG) with no clinically significant abnormalities indicative of myocardial ischemia.
6. Ongoing toxicity associated with prior anticancer therapy ≤ grade 1 Common Terminology Criteria for Adverse Events (CTCAE version 4.03) with the exception of alopecia.
7. Maximum of three prior chemotherapy lines for advanced breast cancer (not including neo/adjuvant chemotherapy). If prior treatment with paclitaxel, PD must have occurred > 12 months from the end of previous adjuvant treatment or for previous metastatic treatment no PD must have occurred during treatment or within 3 months of the end of treatment
8. Life expectancy of at least three months.
9. Patients must be able to swallow and retain oral medication (intact tablet).
10. Able to undergo all screening assessments outlined in the protocol following written informed consent.
11. Adequate organ function (defined by the following parameters):

    1. Serum creatinine < 140 µmol/L or creatinine clearance > 60 mL/min.
    2. Serum hemoglobin ≥ 9 g/dL; absolute neutrophil count ≥ 1.5 x 10**9/L; platelets ≥ 100 x 10**9/L.
    3. Serum bilirubin ≤ 1.5 x upper normal limit (UNL).
    4. Serum ALT, AST ≤ 2.5 x UNL but ≤ 5.0 x UNL in case of liver metastases; ALP ≤ UNL but ≤ 1.5 x ULN in case of liver metastases; albumin within normal limits. If ALP is greater than 1.5 x UNL (in the presence of liver metastases) the liver isoenzyme fraction will be measured. Liver isoenzyme fraction (absolute value) must be ≤ 1.5 x UNL.
12. No known hepatitis B virus (not due to immunization), hepatitis C virus, human immunodeficiency virus Ι and -ΙΙ positive status.

Exclusion Criteria:

1. Male.
2. Pregnancy or lactation or unwillingness to use adequate method of birth control.
3. HER-2 positive disease status.
4. Less than four weeks since last chemotherapy, radiotherapy or prior investigational therapy. Less than two weeks since last hormone or immunotherapy or signal transduction therapy.
5. Neurological or psychiatric disorders which may influence understanding of study and informed consent procedures.
6. Active or uncontrolled infection.
7. Malabsorption syndrome, disease significantly affecting gastrointestinal function.
8. Hypersensitivity to:

   1. paclitaxel
   2. ibuprofen or to more than one non-steroidal anti-inflammatory drug.
   3. medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib.
9. Presence of brain metastases (this does not include primary brain tumors) or leptomeningeal disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2014-06-25 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, MD, Principal Investigator — University of Michigan; Lori Goldstein, MD, Principal Investigator — Fox Chase Cancer Center; Raymond Perez, MD, Principal Investigator — University of Kansas Medical Center; Tiffany Avery, MD, Principal Investigator — Thomas Jefferson University; Giraldo Kato, MD, Principal Investigator — Pinnacle Oncology Hematology
Locations (5):
- United States (5):
  - Pinnacle Oncology Hematology; 9055 East Del Camino, Scottsdale, Arizona
  - University of Kansas Medical Center; 4350 Shawnee Mission Parkway, Fairway, Kansas
  - University of Michigan; 1500 East Medical Center Drive, Ann Arbor, Michigan
  - Thomas Jefferson University Hospital; 1025 Walnut Street, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center; 333 Cottman Avenue, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pts were enrolled in a staggered way. 1 pt was enrolled; if no Dose Limiting Toxicity (DLT) was observed by Day 8, 2 further pts were enrolled simultaneously. If no DLTs were observed at the end of 1 cycle, escalation to the next dose was considered and hence, 3 further pts were enrolled simultaneously. After reviewing Cycle 1 data, escalation to the next dose level was considered. Escalation was stopped if 2 pts of the initial 3 or the expanded cohort of 6 pts developed DLTs.
Pre-assignment Details: Reparixin + paclitaxel were administered in 28-day cycles as long as clinical benefit was observed.
  Reparixin was administered in oral tablets every six to ten hours during a 3 day run-in period and for 21 consecutive days during each cycle with 7 days off treatment between each cycle.
  Paclitaxel 80 mg/m2/week was administered in combination with the day's first dose of reparixin as an i.v. infusion on Days 1, 8 and 15 of each 28-day cycle.
Groups:
- Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 400 mg t.i.d.; Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 800 mg t.i.d.: Paclitaxel+reparixin three weeks on one week off (three to six patients)
  Paclitaxel+Reparixin: Association of Paclitaxel at fixed dosage with three increasing dosage of Reparixin
- Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 1200 mg t.i.d.: Paclitaxel+reparixin oral three weeks on one week off (three to six patients).
  Paclitaxel+Reparixin: Association of Paclitaxel at fixed dosage with three increasing dosage of Reparixin
Period: Run-in Period
Arm/Group | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 400 mg t.i.d. | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 800 mg t.i.d. | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 1200 mg t.i.d.
Started | 4 | 3 | 26
Completed | 4 | 3 | 26
Not Completed | 0 | 0 | 0
Period: Reparixin + Paclitaxel (28-day Cycles)
Arm/Group | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 400 mg t.i.d. | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 800 mg t.i.d. | Paclitaxel 80 mg/m2 i.v.+Reparixin Oral 1200 mg t.i.d.
Started | 4 | 3 | 26
Completed | 0 | 0 | 0
Not Completed | 4 | 3 | 26
Not completed — Disease progression | 2 | 3 | 14
Not completed — Adverse Event | 1 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 4 | 3 | 23 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 16 | 22
  >=65 years | 1 | 0 | 7 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.13) | 55.3 (7.77) | 56.2 (12.69) | 55.9 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 23 | 30
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 22 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 3 | 1 | 20 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 23 | 30

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Events (TEAEs)
Description: Monitoring of AEs throughout the study till the end/off-treatment visit.
Time Frame: Up to 28 days following the last dose of study drug (up to 24 months).
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Number; unit: adverse events
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
adverse events | 106 | 99 | 506

2. Primary Outcome: Plasma DF1681Y Concentrations by Time Point
Description: Plasma DF 1681Y concentrations are reported by time point for the PK Population. The CSR also presents:
  * plots of mean plasma PK concentrations versus time for DF 1681Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population;
  * plots of individual plasma PK concentrations versus time for DF 1681Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population; and
  * a plot of reparixin versus time on Day -3 and Day 21 on a linear (upper) or semi-log (lower) axis.
Time Frame: Days -3 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours), 1 (0, 0.5, 1, 2, 4, 8, 24 hours), 8 (0, 0.5, 1, 2, 4, 8, 24 hours), and 21 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours) of cycle 1.
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Day -3 - 0 hr | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Day -3 - 0.5 hr | 20.648 (22.1597) | 25.743 (25.4196) | 34.689 (34.8550)
  Day -3 - 1 hr | 27.683 (19.5342) | 26.780 (28.4543) | 48.653 (27.4858)
  Day -3 - 1.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day -3 - 1.5 hr | 31.038 (15.2190) | 22.180 (14.3448) | 55.810 (22.6579)
  Day -3 - 2 hr | 22.020 (11.0967) | 20.253 (12.2131) | 50.630 (17.8120)
  Day -3 - 3 hr | 12.868 (5.8392) | 18.650 (8.4463) | 30.968 (10.7100)
  Day -3 - 4 hr | 8.233 (4.9883) | 14.933 (7.2954) | 20.747 (8.4992)
  Day -3 - 6 hr | 2.838 (2.1480) | 6.537 (2.6240) | 9.650 (7.3114)
  Day -3 - 8 hr | 1.538 (0.6268) | 3.980 (2.1701) | 8.768 (12.3086)
  Day 1 - 0 hr | 1.050 (0.3705) | 4.243 (3.3862) | 5.739 (6.7727)
  Day 1 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0.5 hr | 21.503 (22.1075) | 26.023 (16.2351) | 21.407 (23.0450)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 19.553 (19.5114) | 45.413 (3.8760) | 39.378 (31.5133)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 22.420 (13.4937) | 31.090 (10.9918) | 47.519 (21.1919)
  Day 1 - 4 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 4 hr | 9.923 (5.3392) | 11.127 (3.5750) | 27.033 (14.4401)
  Day 1 - 8 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 8 hr | 2.185 (0.8552) | 2.733 (1.1838) | 17.579 (23.5794)
  Day 1 - 24 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 24 hr | 23.667 (31.3613) | 23.193 (13.3628) | 19.685 (21.7424)
  Day 8 - 0 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0 hr | 0.785 (1.0511) | 2.403 (1.7784) | 3.549 (2.0530)
  Day 8 - 0.5 hr: number analyzed (Participants) | 4 | 2 | 10
  Day 8 - 0.5 hr | 8.010 (4.5690) | 5.689 (6.7670) | 38.937 (39.3111)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 14.178 (9.3500) | 21.383 (21.5045) | 35.506 (29.9050)
  Day 8 - 2 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 2 hr | 14.110 (9.4066) | 30.897 (7.7797) | 34.182 (23.7096)
  Day 8 - 4 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 4 hr | 9.360 (6.2105) | 24.717 (6.1212) | 23.986 (15.9604)
  Day 8 - 8 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 8 hr | 2.740 (1.4252) | 7.807 (3.7770) | 11.111 (17.0215)
  Day 8 - 24 hr: number analyzed (Participants) | 4 | 3 | 9
  Day 8 - 24 hr | 22.000 (27.8459) | 14.843 (18.6946) | 10.394 (7.5534)
  Day 21 - 0 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0 hr | 1.247 (0.7580) | 6.003 (5.5644) | 4.978 (4.3227)
  Day 21 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0.5 hr | 2.187 (0.7559) | 29.380 (31.8622) | 48.578 (28.9433)
  Day 21 - 1 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1 hr | 3.883 (1.1319) | 36.397 (33.4112) | 62.916 (28.5967)
  Day 21 - 1.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1.5 hr | 10.113 (5.4962) | 33.787 (25.5501) | 54.749 (19.5782)
  Day 21 - 2 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 2 hr | 13.433 (9.0774) | 29.663 (17.0469) | 43.490 (20.5604)
  Day 21 - 3 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 3 hr | 18.677 (2.3019) | 24.693 (7.9406) | 24.698 (13.4553)
  Day 21 - 4 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 4 hr | 8.897 (2.5150) | 17.780 (2.4222) | 17.359 (10.2954)
  Day 21 - 6 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 6 hr | 3.247 (0.6596) | 12.383 (6.9546) | 7.041 (3.9328)
  Day 21 - 8 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 8 hr | 2.003 (0.2380) | 5.607 (2.1608) | 3.684 (2.2504)

3. Primary Outcome: Plasma Unbound DF1681Y Concentrations by Time Point
Description: Plasma unbound DF 1681Y concentrations by time point for the PK Population are reported. CSR also presents:
  * plots of mean plasma PK concentrations versus time for unbound DF 1681Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population; and
  * plots of individual plasma PK concentrations versus time for unbound DF 1681Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population.
Time Frame: Days -3 (1, 2 hours), 1 (1, 2 hours), 8 (1, 2 hours), and 21 (1, 2 hours) of cycle 1.
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ng/mL
  Day -3 - 1 hr | 13.7 (10.13) | 22.4 (19.14) | 109.1 (131.15)
  Day -3 - 2 hr | 13.1 (7.27) | 37.2 (26.35) | 74.5 (63.82)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 12.3 (14.64) | 78.9 (38.86) | 76.2 (107.84)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 13.2 (7.79) | 25.0 (11.57) | 83.9 (97.73)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 9.1 (7.63) | 13.0 (13.27) | 84.4 (147.04)
  Day 8 - 2 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 2 hr | 9.3 (5.00) | 21.6 (8.37) | 30.4 (29.46)
  Day 21 - 1 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1 hr | 2.5 (0.96) | 44.9 (61.18) | 117.2 (84.65)
  Day 21 - 2 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 2 hr | 14.9 (16.49) | 34.1 (21.54) | 50.8 (42.04)

4. Primary Outcome: Plasma DF2243Y Concentrations by Time Point
Description: DF2243Y, DF2188Y, methanesulfonamide and ibuprofen are the metabolites detected in human plasma and urine, with DF2243Y being the major metabolite. Plasma DF 2243Y concentrations by time point for the PK Population are reported. CSR also presents:
  * plots of mean plasma PK concentrations versus time for DF 2243Y on Days -3, 1, 8 and 21, respectively (linear and semi-logarithmic) for the PK Population;
  * plots of individual plasma PK concentrations versus time for DF 2243Y on Days -3, 1, 8 and 21 (linear and semi-logarithmic) for the PK Population;
  * a plot of DF 2243Y versus time on Day -3 and Day 21 on a linear (upper) or semi-log (lower) axis.
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Day -3 - 0 hr | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day -3 - 0.5 hr | 0.188 (0.1477) | 0.167 (0.1943) | 0.813 (1.2689)
  Day -3 - 1 hr | 0.905 (0.4641) | 1.380 (1.6229) | 4.679 (4.8768)
  Day -3 - 1.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day -3 - 1.5 hr | 2.760 (1.5317) | 2.803 (2.3608) | 10.339 (7.9404)
  Day -3 - 2 hr | 4.990 (2.2479) | 4.470 (2.7070) | 14.382 (7.8212)
  Day -3 - 3 hr | 5.478 (1.6318) | 7.497 (4.2183) | 18.168 (7.3720)
  Day -3 - 4 hr | 4.743 (0.1638) | 7.857 (3.7009) | 16.806 (5.3131)
  Day -3 - 6 hr | 2.753 (1.1919) | 6.000 (0.6744) | 11.187 (4.8182)
  Day -3 - 8 hr | 1.660 (1.1473) | 3.693 (1.1453) | 6.935 (4.18711)
  Day 1 - 0 hr | 1.078 (0.5890) | 4.683 (5.2831) | 6.524 (7.2445)
  Day 1 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0.5 hr | 1.008 (0.4421) | 4.987 (4.8793) | 5.878 (6.5607)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 2.023 (0.0645) | 6.520 (4.1584) | 7.027 (6.0291)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 4.218 (2.0817) | 13.093 (4.0594) | 14.229 (8.7457)
  Day 1 - 4 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 4 hr | 5.228 (2.7555) | 11.727 (1.3886) | 19.320 (8.1202)
  Day 1 - 8 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 8 hr | 1.555 (0.5630) | 2.933 (0.4864) | 11.402 (8.7268)
  Day 1 - 24 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 24 hr | 5.507 (4.0277) | 12.953 (7.3222) | 12.365 (10.8597)
  Day 8 - 0 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0 hr | 0.768 (0.8572) | 2.787 (2.6405) | 6.435 (7.0355)
  Day 8 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0.5 hr | 0.710 (0.7590) | 2.595 (2.9911) | 5.927 (4.2413)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 1.118 (0.8848) | 2.850 (2.2700) | 8.123 (5.8406)
  Day 8 - 2 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 2 hr | 3.873 (3.7232) | 6.080 (3.6576) | 16.459 (10.0027)
  Day 8 - 4 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 4 hr | 6.447 (3.9722) | 9.960 (1.3869) | 16.595 (6.9212)
  Day 8 - 8 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 8 hr | 2.080 (0.4491) | 4.320 (1.1801) | 8.401 (6.9080)
  Day 8 - 24 hr: number analyzed (Participants) | 2 | 3 | 9
  Day 8 - 24 hr | 4.205 (1.5768) | 3.310 (1.3343) | 10.500 (8.1986)
  Day 21 - 0 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0 hr | 2.090 (2.2439) | 3.923 (3.1708) | 5.984 (4.0332)
  Day 21 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0.5 hr | 1.373 (1.1150) | 3.577 (2.9258) | 5.833 (3.6968)
  Day 21 - 1 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1 hr | 1.593 (1.1089) | 5.650 (5.6922) | 11.106 (7.6876)
  Day 21 - 1.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1.5 hr | 1.777 (1.0633) | 7.097 (7.0797) | 15.220 (7.9701)
  Day 21 - 2 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 2 hr | 2.333 (1.4514) | 8.093 (6.9801) | 19.603 (9.6539)
  Day 21 - 3 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 3 hr | 5.650 (2.3079) | 10.343 (5.5662) | 18.900 (8.1250)
  Day 21 - 4 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 4 hr | 7.320 (1.7217) | 8.947 (3.6574) | 16.361 (6.5721)
  Day 21 - 6 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 6 hr | 4.090 (0.9231) | 7.597 (3.2853) | 11.146 (5.9542)
  Day 21 - 8 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 8 hr | 2.070 (0.3811) | 4.497 (1.9566) | 7.086 (5.3867)

5. Primary Outcome: Plasma DF2188Y Concentrations by Time Point
Description: DF2243Y, DF2188Y, methanesulfonamide and ibuprofen are the metabolites detected in human plasma and urine, with DF2243Y being the major metabolite. Plasma DF 2188Y concentrations by time point for the PK Population are reported. CSR also presents:
  * a plot of mean plasma PK concentrations versus time for DF 2188Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population;
  * plots of individual plasma PK concentrations versus time for DF 2188Y on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population;
  * a plot of DF 2881Y versus time on Day -3 and Day 21 on a linear (upper) or semi-log (lower) axis.
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Day -3 - 0 hr | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day -3 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 12
  Day -3 - 0.5 hr | 0.547 (0.3798) | 0.717 (0.8503) | 1.781 (2.4828)
  Day -3 - 1 hr | 1.311 (0.6671) | 2.128 (2.3765) | 4.986 (3.6296)
  Day -3 - 1.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day -3 - 1.5 hr | 2.337 (0.9274) | 2.581 (2.0086) | 8.136 (3.7429)
  Day -3 - 2 hr | 2.882 (1.1328) | 2.693 (1.0611) | 9.381 (5.0573)
  Day -3 - 3 hr | 2.024 (0.4877) | 2.968 (1.0848) | 8.332 (4.3300)
  Day -3 - 4 hr | 1.455 (0.5505) | 2.752 (0.5639) | 5.320 (2.8278)
  Day -3 - 6 hr | 0.571 (0.2527) | 1.732 (0.4955) | 2.373 (1.2315)
  Day -3 - 8 hr | 0.385 (0.2775) | 0.891 (0.4059) | 1.813 (1.5823)
  Day 1 - 0 hr | 0.243 (0.1092) | 1.360 (1.7820) | 1.433 (2.0366)
  Day 1 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0.5 hr | 0.997 (0.4469) | 2.930 (0.9101) | 2.324 (2.7844)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 1.883 (1.0503) | 7.251 (1.4929) | 6.940 (6.5771)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 2.804 (1.5570) | 6.129 (0.5653) | 12.093 (8.5639)
  Day 1 - 4 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 4 hr | 1.687 (0.7018) | 3.103 (0.6448) | 8.951 (6.3792)
  Day 1 - 8 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 8 hr | 0.342 (0.1840) | 0.519 (0.2349) | 4.222 (3.8268)
  Day 1 - 24 hr: number analyzed (Participants) | 3 | 3 | 11
  Day 1 - 24 hr | 2.019 (1.8027) | 4.706 (2.4979) | 5.249 (7.1068)
  Day 8 - 0 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0 hr | 0.185 (0.2617) | 0.536 (0.4428) | 1.302 (1.9543)
  Day 8 - 0.5 hr: number analyzed (Participants) | 4 | 2 | 10
  Day 8 - 0.5 hr | 0.381 (0.2595) | 0.913 (1.1455) | 7.260 (9.2883)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 1.360 (1.0877) | 2.022 (1.5295) | 9.494 (8.6619)
  Day 8 - 2 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 2 hr | 2.159 (0.9085) | 4.423 (0.8932) | 10.592 (9.1860)
  Day 8 - 4 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 4 hr | 1.966 (1.2606) | 3.552 (0.6505) | 6.181 (3.1973)
  Day 8 - 8 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 8 hr | 0.614 (0.4115) | 1.117 (0.5547) | 2.101 (2.1855)
  Day 8 - 24 hr: number analyzed (Participants) | 2 | 3 | 9
  Day 8 - 24 hr | 1.961 (1.5761) | 1.627 (1.1583) | 2.753 (2.7020)
  Day 21 - 0 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0 hr | 0.348 (0.2480) | 0.913 (0.7577) | 1.211 (1.0054)
  Day 21 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0.5 hr | 0.331 (0.0515) | 1.542 (1.5637) | 3.707 (2.8351)
  Day 21 - 1 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1 hr | 0.398 (0.0494) | 3.039 (3.1614) | 8.087 (4.2863)
  Day 21 - 1.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1.5 hr | 0.911 (0.3382) | 3.522 (2.8731) | 9.590 (4.4184)
  Day 21 - 2 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 2 hr | 1.612 (0.7290) | 3.647 (2.0369) | 9.485 (6.1568)
  Day 21 - 3 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 3 hr | 3.138 (0.9689) | 3982 (1.2720) | 6.382 (4.5496)
  Day 21 - 4 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 4 hr | 2.389 (0.1047) | 3.518 (1.4208) | 4.209 (2.0152)
  Day 21 - 6 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 6 hr | 0.949 (0.1443) | 2.185 (1.2816) | 2.139 (1.9283)
  Day 21 - 8 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 8 hr | 0.482 (0.1344) | 0.987 (0.4603) | 1.166 (1.4547)

6. Primary Outcome: Plasma Ibuprofen Concentrations by Time Point
Description: DF2243Y, DF2188Y, methanesulfonamide and ibuprofen are the metabolites detected in human plasma and urine, with DF2243Y being the major metabolite.
  Plasma ibuprofen concentrations are reported by time point for the PK Population. CSR describes also:
  * a plot of mean plasma PK concentrations versus time for ibuprofen on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population;
  * plots of individual plasma PK concentrations versus time for ibuprofen on Days -3, 1, 8 and 21 respectively (linear and semi-logarithmic) for the PK Population;
  * a plot of ibuprofen versus time on Day -3 and Day 21 on a linear (upper) or semi-log (lower) axis.
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Day -3 - 0 hr | 0.040 (0.0383) | 0.024 (0.0172) | 0.030 (0.0444)
  Day -3 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 12
  Day -3 - 0.5 hr | 0.165 (0.1401) | 0.260 (0.3355) | 0.282 (0.2943)
  Day -3 - 1 hr | 0.244 (0.3003) | 0.578 (0.7653) | 1.141 (0.9977)
  Day -3 - 1.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day -3 - 1.5 hr | 0.430 (0.4382) | 0.663 (0.8429) | 2.144 (1.6461)
  Day -3 - 2 hr | 0.676 (0.6193) | 0.736 (0.7971) | 2.728 (2.5583)
  Day -3 - 3 hr | 0.760 (0.6860) | 0.863 (0.6598) | 2.979 (2.6527)
  Day -3 - 4 hr | 0.732 (0.6436) | 0.930 (0.5859) | 2.420 (2.3095)
  Day -3 - 6 hr | 0.564 (0.5032) | 0.861 (0.5131) | 1.653 (1.3698)
  Day -3 - 8 hr | 0.453 (0.3960) | 0.680 (0.4165) | 1.249 (0.9589)
  Day 1 - 0 hr | 0.414 (0.4035) | 1.245 (1.3888) | 1.077 (0.9690)
  Day 1 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0.5 hr | 0.410 (0.3334) | 1.2220 (1.0325) | 0.984 (0.8270)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 0.539 (0.5508) | 1.759 (1.5027) | 1.319 (1.2569)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 0.798 (0.8648) | 1.948 (1.4572) | 2.633 (2.2699)
  Day 1 - 4 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 4 hr | 0.816 (0.8769) | 1.557 (0.9902) | 2.575 (2.0191)
  Day 1 - 8 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 8 hr | 0.440 (0.3806) | 0.693 (0.4651) | 1.532 (1.0465)
  Day 1 - 24 hr: number analyzed (Participants) | 3 | 3 | 11
  Day 1 - 24 hr | 0.862 (0.4607) | 1.964 (1.5247) | 1.667 (1.3126)
  Day 8 - 0 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0 hr | 0.125 (0.1307) | 0.534 (0.5566) | 1.068 (0.7676)
  Day 8 - 0.5 hr: number analyzed (Participants) | 4 | 2 | 10
  Day 8 - 0.5 hr | 0.140 (0.1191) | 0.652 (0.7177) | 2.087 (2.0162)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 0.251 (0.2304) | 0.571 (0.5765) | 2.683 (2.7211)
  Day 8 - 2 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 2 hr | 0.312 (0.3725) | 1.065 (0.8626) | 2.879 (2.7853)
  Day 8 - 4 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 4 hr | 0.352 (0.3909) | 1.016 (0.4036) | 2.553 (2.0585)
  Day 8 - 8 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 8 hr | 0.213 (0.2363) | 0.699 (0.4269) | 1.310 (1.0034)
  Day 8 - 24 hr: number analyzed (Participants) | 2 | 3 | 9
  Day 8 - 24 hr | 0.416 (0.4582) | 0.602 (0.3706) | 1.448 (0.9161)
  Day 21 - 0 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0 hr | 0.300 (0.3560) | 0.863 (0.7528) | 1.210 (0.8951)
  Day 21 - 0.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 0.5 hr | 0.226 (0.2443) | 0.734 (0.5966) | 1.341 (0.7483)
  Day 21 - 1 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1 hr | 0.238 (0.2627) | 0.849 (0.6339) | 2.381 (1.4899)
  Day 21 - 1.5 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 1.5 hr | 0.237 (0.2291) | 0.986 (0.7064) | 3.222 (2.2855)
  Day 21 - 2 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 2 hr | 0.342 (0.3656) | 1.214 (0.8686) | 3.335 (2.4454)
  Day 21 - 3 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 3 hr | 0.543 (0.5866) | 1.562 (1.1380) | 3.327 (2.8221)
  Day 21 - 4 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 4 hr | 0.546 (0.6712) | 1.970 (1.9069) | 2.712 (1.9665)
  Day 21 - 6 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 6 hr | 0.404 (0.4958) | 1.179 (0.6063) | 1.645 (1.2753)
  Day 21 - 8 hr: number analyzed (Participants) | 3 | 3 | 9
  Day 21 - 8 hr | 0.312 (0.227) | 0.802 (0.3472) | 1.218 (0.9901)

7. Primary Outcome: Plasma Paclitaxel Concentrations by Time Point
Description: Plasma paclitaxel concentrations are reported by time point for the PK Population. CSR describes also:
  * A plot of mean plasma PK concentrations versus time for paclitaxel on Days 1 and 8 respectively (linear and semi-logarithmic) for the PK Population;
  * plots of individual plasma PK concentrations versus time for paclitaxel on Days 1 and 8 respectively (linear and semi-logarithmic) for the PK Population;
  * a plot of paclitaxel versus time on Day 1 and Day 8 on a linear (upper) or semi-log (lower) axis.
Time Frame: Days 1 (0, 0.5, 1, 2, 4, 8, 24 hours) and 8 (0, 0.5, 1, 2, 4, 8, 24 hours) of cycle 1.
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Day 1 - 0 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0 hr | 0.000 (0.0000) | 0.000 (0.0000) | 0.070 (0.1664)
  Day 1 - 0.5 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 0.5 hr | 1.483 (1.0948) | 1.560 (0.5060) | 2.275 (1.2319)
  Day 1 - 1 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 1 hr | 1.954 (1.0995) | 2.438 (0.4045) | 2.898 (1.4819)
  Day 1 - 2 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 2 hr | 0.733 (0.7148) | 0.342 (0.1071) | 0.600 (0.4058)
  Day 1 - 4 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 4 hr | 0.166 (0.0560) | 0.118 (0.0398) | 0.363 (0.5901)
  Day 1 - 8 hr: number analyzed (Participants) | 4 | 3 | 11
  Day 1 - 8 hr | 0.066 (0.0094) | 0.060 (0.0190) | 0.099 (0.0622)
  Day 1 - 24 hr: number analyzed (Participants) | 3 | 3 | 11
  Day 1 - 24 hr | 0.019 (0.0076) | 0.020 (0.0076) | 0.030 (0.0145)
  Day 8 - 0 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 0 hr | 0.000 (0.0000) | 0.004 (0.0075) | 0.001 (0.0022)
  Day 8 - 0.5 hr: number analyzed (Participants) | 4 | 2 | 10
  Day 8 - 0.5 hr | 1.409 (1.0059) | 1.466 (0.1372) | 2.426 (1.3387)
  Day 8 - 1 hr: number analyzed (Participants) | 4 | 3 | 10
  Day 8 - 1 hr | 1.730 (1.1795) | 2.554 (0.7296) | 3.222 (1.4919)
  Day 8 - 2 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 2 hr | 0.318 (0.0707) | 0.706 (0.7383) | 0.759 (1.0239)
  Day 8 - 4 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 4 hr | 0.122 (0.0294) | 0.175 (0.1054) | 0.196 (0.1234)
  Day 8 - 8 hr: number analyzed (Participants) | 3 | 3 | 10
  Day 8 - 8 hr | 0.060 (0.0195) | 0.102 (0.0814) | 0.095 (0.0638)
  Day 8 - 24 hr: number analyzed (Participants) | 2 | 3 | 9
  Day 8 - 24 hr | 0.023 (0.0078) | 0.047 (0.0430) | 0.031 (0.0190)

8. Primary Outcome: C0 and Cmax for DF1681Y
Description: PK parameters were calculated for cycle 1 only.
  Co is the pre-dose concentration/concentration at time zero. Cmax is the maximum plasma concentration obtained directly from the data without interpolation, expressed in concentration units.
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  DF1681Y - C0 - Day -3 | 0.00 (0) | 0.00 (0) | 0.00 (0)
  DF1681Y - C0 - Day 1 | 1.05 (0.37) | 4.24 (3.39) | 5.74 (6.77)
  DF1681Y - C0 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF1681Y - C0 - Day 8 | 0.79 (1.05) | 2.40 (1.78) | 3.55 (2.05)
  DF1681Y - C0 - Day 21: number analyzed (Participants) | 3 | 3 | 9
  DF1681Y - C0 - Day 21 | 1.25 (0.76) | 6.00 (5.56) | 4.98 (4.32)
  DF1681Y - Cmax - Day -3 | 37.9 (15.2) | 35.6 (328.6) | 65.0 (21.1)
  DF1681Y - Cmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF1681Y - Cmax - Day 1 | 30.7 (19.0) | 45.4 (3.88) | 58.7 (22.9)
  DF1681Y - Cmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF1681Y - Cmax - Day 8 | 17.9 (7.11) | 34.4 (11.5) | 60.2 (26.5)
  DF1681Y - Cmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF1681Y - Cmax - Day 21 | 19.4 (3.27) | 44.6 (25.3) | 71.2 (24.6)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; DF1681Y Cmax at Day -3; Test type: Other; p = 0.0341, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; DF1681Y Cmax at Day -3; Test type: Other; p = 0.0636, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; DF1681Y Cmax at Day 1; Test type: Other; p = 0.0487, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; DF1681Y Cmax at Day 1; Test type: Other; p = 0.3498, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; DF1681Y Cmax at Day 8; Test type: Other; p = 0.0096, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; DF1681Y Cmax at Day 8; Test type: Other; p = 0.1374, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; DF1681Y Cmax at Day 21; Test type: Other; p = 0.0065, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; DF1681Y Cmax at Day 21; Test type: Other; p = 0.1470, ANOVA

9. Primary Outcome: C0 and Cmax for DF2243Y
Description: as for outcome 8
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  DF2243Y - C0 - Day -3 | 0.00 (0) | 0.00 (0) | 0.00 (0)
  DF2243Y - C0 - Day 1 | 1.08 (0.59) | 4.68 (5.28) | 6.52 (7.25)
  DF2243Y - C0 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2243Y - C0 - Day 8 | 0.77 (0.86) | 2.79 (2.64) | 6.44 (7.04)
  DF2243Y - C0 - Day 21: number analyzed (Participants) | 3 | 3 | 9
  DF2243Y - C0 - Day 21 | 2.09 (2.24) | 3.92 (3.17) | 5.98 (4.03)
  DF2243Y - Cmax - Day -3 | 5.85 (1.50) | 8.46 (3.05) | 19.5 (6.73)
  DF2243Y - Cmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2243Y - Cmax - Day 1 | 5.79 (2.84) | 13.8 (3.51) | 20.6 (8.35)
  DF2243Y - Cmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2243Y - Cmax - Day 8 | 5.07 (4.32) | 10.6 (0.32) | 18.3 (8.22)
  DF2243Y - Cmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2243Y - Cmax - Day 21 | 7.71 (1.63) | 12.6 (3.13) | 21.4 (8.75)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; DF2243 Cmax at Day -3; Test type: Other; p = 0.0015, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; DF2243 Cmax at Day -3; Test type: Other; p = 0.0176, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; DF2243 Cmax at Day 1; Test type: Other; p = 0.0048, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; DF2243 Cmax at Day 1; Test type: Other; p = 0.2083, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 2; DF2243 Cmax at Day 8; Test type: Other; p = 0.0111, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; DF2243 Cmax at Day 8; Test type: Other; p = 0.1441, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; DF2243 Cmax at Day 21; Test type: Other; p = 0.0283, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; DF2243 Cmax at Day 21; Test type: Other; p = 0.1331, ANOVA

10. Primary Outcome: C0 and Cmax for DF2188Y
Description: as for outcome 8
Time Frame: Days -3 (pre-dose, 0.5, 1, 2, 4, 8, 24 hours), 1 (pre-dose, 0.5, 1, 2, 4, 8, 24 hours), 8 (pre-dose, 0.5, 1, 2, 4, 8, 24 hours) and 21 (pre-dose, 0.5, 1, 2, 4, 8, 24 hours)
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  DF2188Y- C0 - Day -3 | 0 (0) | 0 (0) | 0 (0)
  DF2188Y - C0 - Day 1 | 0.24 (0.11) | 1.36 (1.78) | 1.43 (2.04)
  DF2188Y - C0 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2188Y - C0 - Day 8 | 0.18 (0.26) | 0.54 (0.44) | 1.30 (1.95)
  DF2188Y - C0 - Day 21: number analyzed (Participants) | 3 | 3 | 9
  DF2188Y - C0 - Day 21 | 0.35 (0.25) | 0.91 (0.76) | 1.21 (1.01)
  DF2188Y - Cmax - Day -3 | 3.01 (0.99) | 3.67 (1.42) | 10.5 (4.85)
  DF2188Y - Cmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2188Y - Cmax - Day 1 | 2.90 (1.53) | 7.37 (1.29) | 13.4 (7.68)
  DF2188Y - Cmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2188Y - Cmax - Day 8 | 2.11 (1.25) | 4.42 (0.89) | 14.5 (9.30)
  DF2188Y - Cmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2188Y - Cmax - Day 21 | 3.29 (0.73) | 5.27 (2.42) | 12.2 (5.83)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; DF2188Y, Cmax, Day -3; Test type: Other; p = 0.0097, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; DF2188Y, Cmax, Day -3; Test type: Other; p = 0.0354, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; DF2188Y, Cmax, Day 1; Test type: Other; p = 0.0200, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; DF2188Y, Cmax, Day 1; Test type: Other; p = 0.2134, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; DF2188Y, Cmax, Day 8; Test type: Other; p = 0.0235, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; DF2188Y, Cmax, Day 8; Test type: Other; p = 0.0964, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; DF2188Y, Cmax, Day 21; Test type: Other; p = 0.0314, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; DF2188Y, Cmax, Day 21; Test type: Other; p = 0.0773, ANOVA

11. Primary Outcome: C0 and Cmax for Ibuprofen
Description: as for outcome 8
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  ibuprofen - C0 - Day -3 | 0.04 (0.04) | 0.02 (0.02) | 0.03 (0.04)
  ibuprofen - C0 - Day 1 | 0.41 (0.40) | 1.25 (1.39) | 1.08 (0.97)
  ibuprofen - C0 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  ibuprofen - C0 - Day 8 | 0.12 (0.13) | 0.53 (0.56) | 1.07 (0.77)
  ibuprofen - C0 - Day 21: number analyzed (Participants) | 3 | 3 | 9
  ibuprofen - C0 - Day 21 | 0.3 (0.36) | 0.86 (0.75) | 1.21 (0.90)
  ibuprofen - Cmax - Day -3: number analyzed (Participants) | 4 | 3 | 9
  ibuprofen - Cmax - Day -3 | 0.77 (0.78) | 1.02 (0.59) | 3.11 (2.59)
  ibuprofen - Cmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  ibuprofen - Cmax - Day 1 | 0.86 (0.86) | 1.98 (1.46) | 2.95 (2.10)
  ibuprofen - Cmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  ibuprofen - Cmax - Day 8 | 0.34 (0.32) | 1.24 (0.75) | 3.69 (2.67)
  ibuprofen - Cmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  ibuprofen - Cmax - Day 21 | 0.58 (0.64) | 2.16 (1.74) | 3.99 (2.74)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Cmax, ibuprofen, Day -3; Test type: Other; p = 0.1016, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day -3; Test type: Other; p = 0.2001, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; Cmax, ibuprofen, Day 1; Test type: Other; p = 0.0802, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day 1; Test type: Other; p = 0.4728, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; Cmax, ibuprofen, Day 8; Test type: Other; p = 0.0355, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day 8; Test type: Other; p = 0.1709, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Cmax, ibuprofen, Day 21; Test type: Other; p = 0.0685, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day 21; Test type: Other; p = 0.3189, ANOVA

12. Primary Outcome: Cmax for Paclitaxel
Description: as for outcome 8
Time Frame: Days 1 (0, 0.5, 1, 2, 4, 8, 24 hours), 8 (0, 0.5, 1, 2, 4, 8, 24 hours)
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ug/mL
  Paclitaxel - Cmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  Paclitaxel - Cmax - Day 1 | 2.35 (0.47) | 2.44 (0.41) | 3.10 (1.16)
  Paclitaxel - Cmax - Day 8: number analyzed (Participants) | 3 | 3 | 10
  Paclitaxel - Cmax - Day 8 | 2.31 (0.30) | 2.55 (0.73) | 3.62 (0.96)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Paclitaxel, Cmax, Day 1; Test type: Other; p = 0.2375, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day 1; Test type: Other; p = 0.3608, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; Cmax, ibuprofen, Day 8; Test type: Other; p = 0.0442, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; Cmax, ibuprofen, Day 8; Test type: Other; p = 0.1067, ANOVA

13. Primary Outcome: Tmax and t1/2 for DF1681Y
Description: PK parameters were calculated for cycle 1 only. Tmax is the Time to reach the maximum plasma concentration obtained directly from the data without interpolation.
  t1/2 is the Elimination half-life, calculated as ln(2)/ Kel (where Kel is the Terminal elimination rate constant, calculated as the negative of the slope of the terminal log-linear segment of the plasma concentration time curve).
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hours
  DF1681Y - tmax - Day -3 | 0.90 (0.45) | 1.82 (1.25) | 1.41 (0.55)
  DF1681Y - tmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF1681Y - tmax - Day 1 | 2.15 (1.44) | 1.01 (0.01) | 2.64 (4.07)
  DF1681Y - tmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF1681Y - tmax - Day 8 | 1.30 (0.46) | 1.72 (0.48) | 2.45 (2.35)
  DF1681Y - tmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF1681Y - tmax - Day 21 | 2.66 (0.57) | 2.32 (1.52) | 1.40 (0.35)
  DF1681Y - t1/2 - Day -3: number analyzed (Participants) | 4 | 2 | 11
  DF1681Y - t1/2 - Day -3 | 1.65 (0.51) | 1.82 (0.82) | 1.91 (0.64)
  DF1681Y - t1/2 - Day 1: number analyzed (Participants) | 1 | 3 | 3
  DF1681Y - t1/2 - Day 1 | 1.97 | 1.73 (0.09) | 2.14 (0.45)
  DF1681Y - t1/2 - Day 8: number analyzed (Participants) | 1 | 1 | 4
  DF1681Y - t1/2 - Day 8 | 2.00 | 3.57 | 1.88 (0.27)
  DF1681Y - t1/2 - Day 21: number analyzed (Participants) | 2 | 2 | 8
  DF1681Y - t1/2 - Day 21 | 1.89 (0.57) | 1.97 (0.55) | 1.95 (0.56)

14. Primary Outcome: Tmax and t1/2 for DF2243Y
Description: as for outcome 13
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hours
  DF2243Y - tmax - Day -3 | 3.30 (0.87) | 4.32 (1.52) | 3.41 (1.00)
  DF2243Y - tmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2243Y - tmax - Day 1 | 3.51 (0.99) | 2.67 (1.16) | 4.00 (1.57)
  DF2243Y - tmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2243Y - tmax - Day 8 | 4.29 (2.94) | 3.32 (1.15) | 3.40 (1.90)
  DF2243Y - tmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2243Y - tmax - Day 21 | 3.71 (0.62) | 3.66 (2.08) | 2.87 (0.83)
  DF2243Y - t1/2 - Day -3: number analyzed (Participants) | 1 | 1 | 7
  DF2243Y - t1/2 - Day -3 | 1.34 | 3.79 | 2.81 (1.20)
  DF2243Y - t1/2 - Day 1: number analyzed (Participants) | 0 | 0 | 0
  DF2243Y - t1/2 - Day 8: number analyzed (Participants) | 0 | 0 | 0
  DF2243Y - t1/2 - Day 21: number analyzed (Participants) | 1 | 2 | 6
  DF2243Y - t1/2 - Day 21 | 1.97 | 2.46 (0.59) | 3.35 (1.63)

15. Primary Outcome: Tmax and t1/2 for DF2188Y
Description: as for outcome 13
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hours
  DF2188Y - tmax - Day -3 | 2.05 (0.71) | 2.81 (1.24) | 2.44 (1.08)
  DF2188Y- tmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2188Y- tmax - Day 1 | 1.78 (0.52) | 1.33 (0.58) | 2.45 (1.04)
  DF2188Y - tmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2188Y - tmax - Day 8 | 2.30 (1.23) | 2.03 (0.06) | 2.20 (1.37)
  DF2188Y - tmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2188Y - tmax - Day 21 | 3.33 (0.57) | 2.33 (1.14) | 1.77 (0.96)
  DF2188Y - t1/2 - Day -3: number analyzed (Participants) | 3 | 2 | 7
  DF2188Y - t1/2 - Day -3 | 1.63 (0.23) | 2.53 (1.53) | 1.65 (0.40)
  DF2188Y - t1/2 - Day 1: number analyzed (Participants) | 1 | 2 | 0
  DF2188Y - t1/2 - Day 1 | 1.51 | 1.48 (0.07) |
  DF2188Y - t1/2 - Day 8: number analyzed (Participants) | 0 | 0 | 3
  DF2188Y - t1/2 - Day 8 |  |  | 1.42 (0.15)
  DF2188Y - t1/2 - Day 21: number analyzed (Participants) | 2 | 2 | 7
  DF2188Y - t1/2 - Day 21 | 1.90 (0.20) | 1.77 (0.21) | 2.18 (1.44)

16. Primary Outcome: Tmax and t1/2 for Ibuprofen
Description: as for outcome 13
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hours
  DF2188Y - tmax - Day -3 | 3.50 (0.58) | 3.99 (1.99) | 2.86 (0.81)
  DF2188Y- tmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2188Y- tmax - Day 1 | 4.02 (2.86) | 2.66 (1.16) | 4.00 (2.18)
  DF2188Y - tmax - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2188Y - tmax - Day 8 | 4.29 (2.94) | 3.32 (1.15) | 2.15 (1.44)
  DF2188Y - tmax - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2188Y - tmax - Day 21 | 3.37 (0.67) | 3.99 (2.00) | 2.58 (0.97)
  DF2188Y - t1/2 - Day -3: number analyzed (Participants) | 2 | 1 | 6
  DF2188Y - t1/2 - Day -3 | 6.76 (2.04) | 6.15 | 3.76 (0.77)
  DF2188Y - t1/2 - Day 1: number analyzed (Participants) | 0 | 0 | 0
  DF2188Y - t1/2 - Day 8: number analyzed (Participants) | 0 | 0 | 2
  DF2188Y - t1/2 - Day 8 |  |  | 2.15 (0.09)
  DF2188Y - t1/2 - Day 21: number analyzed (Participants) | 2 | 1 | 6
  DF2188Y - t1/2 - Day 21 | 3.12 (0.56) | 3.81 | 3.15 (0.53)

17. Primary Outcome: Tmax and t1/2 for Paclitaxel
Description: as for outcome 13
Time Frame: Days 1 (0, 0.5, 1, 2, 4, 8, 24 hours), 8 (0, 0.5, 1, 2, 4, 8, 24 hours)
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hours
  paclitaxel - tmax - Day 1: number analyzed (Participants) | 4 | 3 | 11
  paclitaxel - tmax - Day 1 | 1.14 (0.63) | 1.01 (0.01) | 1.22 (0.93)
  paclitaxel - tmax - Day 8: number analyzed (Participants) | 3 | 3 | 10
  paclitaxel - tmax - Day 8 | 1.06 (0.09) | 1.06 (0.10) | 1.07 (0.36)
  paclitaxel - t1/2 - Day 1: number analyzed (Participants) | 4 | 3 | 10
  paclitaxel - t1/2 - Day 1 | 5.95 (2.66) | 8.51 (0.43) | 8.18 (0.94)
  paclitaxel - t1/2 - Day 8: number analyzed (Participants) | 3 | 3 | 9
  paclitaxel - t1/2 - Day 8 | 6.57 (3.40) | 11.00 (2.21) | 8.76 (1.05)

18. Primary Outcome: AUC0-8 for DF1681Y
Description: PK parameters were calculated for cycle 1 only. AUC0-8 is the area under the plasma concentration-time curve from time 0 to 8 hours post-dose; calculated using the linear trapezoidal method.
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hr*mg/mL
  DF1681Y - AUC0-8 - Day -3 | 86.7 (34.5) | 108 (58.1) | 194 (71.96)
  DF1681Y - AUC0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF1681Y - AUC0-8 - Day 1 | 86.5 (40.3) | 124 (32.2) | 216 (96.91)
  DF1681Y - AUC0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 8
  DF1681Y - AUC0-8 - Day 8 | 49.8 (38.4) | 150 (44.0) | 178 (88.1)
  DF1681Y - AUC0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF1681Y - AUC0-8 - Day 21 | 57.6 (11.8) | 153 (47.2) | 191 (61.6)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; DF1681Y, AUC0-8, Day -3; Test type: Other; p = 0.0134, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; DF1681Y, AUC0-8, Day -3; Test type: Other; p = 0.0799, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; DF1681Y, AUC0-8, Day 1; Test type: Other; p = 0.0241, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; DF1681Y, AUC0-8, Day 1; Test type: Other; p = 0.01384, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; DF1681Y, AUC0-8, Day 8; Test type: Other; p = 0.0091, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; DF1681Y, AUC0-8, Day 8; Test type: Other; p = 0.5687, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; DF1681Y, AUC0-8, Day 21; Test type: Other; p = 0.0058, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; DF1681Y, AUC0-8, Day 21; Test type: Other; p = 0.3667, ANOVA

19. Primary Outcome: AUC0-8 for DF2243Y
Description: as for outcome 18
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hr*mg/mL
  DF2243Y - AUC0-8 - Day -3 | 25.03 (4.05) | 40.4 (11.9) | 90.21 (35.3)
  DF2243Y - AUC0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2243Y - AUC0-8 - Day 1 | 25.8 (9.2) | 65.0 (13.8) | 108.7 (55.2)
  DF2243Y - AUC0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2243Y - AUC0-8 - Day 8 | 21.6 (18.4) | 49.8 (7.89) | 99.0 (53.2)
  DF2243Y - AUC0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2243Y - AUC0-8 - Day 21 | 31.0 (7.50) | 58.1 (17.7) | 108 (50.5)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; DF2243Y - AUC0-8 - Day -3; Test type: Other; p = 0.0029, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; DF2243Y - AUC0-8 - Day -3; Test type: Other; p = 0.0349, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; DF2243Y - AUC0-8 - Day 1; Test type: Other; p = 0.0119, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; DF2243Y - AUC0-8 - Day 1; Test type: Other; p = 0.2100, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; DF2243Y - AUC0-8 - Day 8; Test type: Other; p = 0.0165, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; DF2243Y - AUC0-8 - Day 8; Test type: Other; p = 0.1496, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; DF2243Y - AUC0-8 - Day 21; Test type: Other; p = 0.0321, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; DF2243Y - AUC0-8 - Day 21; Test type: Other; p = 0.1404, ANOVA

20. Primary Outcome: AUC0-8 for DF2188Y
Description: as for outcome 18
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hr*mg/mL
  DF2188Y - AUC0-8 - Day -3 | 9.79 (1.77) | 16.0 (4.54) | 36.3 (16.8)
  DF2188Y - AUC0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2188Y - AUC0-8 - Day 1 | 11.0 (3.93) | 24.6 (0.86) | 57.2 (39.4)
  DF2188Y - AUC0-8 - Day 8: number analyzed (Participants) | 4 | 2 | 10
  DF2188Y - AUC0-8 - Day 8 | 8.2 (6.01) | 20.8 (2.93) | 46.5 (29.0)
  DF2188Y - AUC0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2188Y - AUC0-8 - Day 21 | 11.0 (1.83) | 21.2 (3.56) | 36.6 (21.6)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; AUC0-8 for DF2188Y, Day -3; Test type: Other; p = 0.0081, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; AUC0-8 for DF2188Y, Day -3; Test type: Other; p = 0.0640, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; AUC0-8 for DF2188Y, Day 1; Test type: Other; p = 0.0397, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; AUC0-8 for DF2188Y, Day 1; Test type: Other; p = 0.1898, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; AUC0-8 for DF2188Y, Day 8; Test type: Other; p = 0.0250, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; AUC0-8 for DF2188Y, Day 8; Test type: Other; p = 0.1605, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; AUC0-8 for DF2188Y, Day 21; Test type: Other; p = 0.0786, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; AUC0-8 for DF2188Y, Day 21; Test type: Other; p = 0.2652, ANOVA

21. Primary Outcome: AUC0-8 for Ibuprofen
Description: as for outcome 18
Time Frame: as for outcome 2
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hr*mg/mL
  ibuprofen - AUC0-8 - Day -3 | 4.35 (3.90) | 5.97 (4.38) | 14.8 (12.7)
  ibuprofen - AUC0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  ibuprofen - AUC0-8 - Day 1 | 5.14 (5.21) | 10.93 (7.55) | 16.17 (12.07)
  ibuprofen - AUC0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  ibuprofen - AUC0-8 - Day 8 | 1.69 (2.29) | 6.82 (4.08) | 17.5 (13.8)
  ibuprofen - AUC0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  ibuprofen - AUC0-8 - Day 21 | 3.17 (3.76) | 9.96 (6.75) | 19.4 (13.3)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Ibuprofen, AUC0-8, Day -3; Test type: Other; p = 0.1335, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day -3; Test type: Other; p = 0.2658, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; Ibuprofen, AUC0-8, Day 1; Test type: Other; p = 0.1063, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day 1; Test type: Other; p = 0.4959, ANOVA
Statistical Analysis 5: Comparison: Group 1 vs Group 3; Ibuprofen, AUC0-8, Day 8; Test type: Other; p = 0.0452, ANOVA
Statistical Analysis 6: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day 8; Test type: Other; p = 0.2223, ANOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 3; Ibuprofen, AUC0-8, Day 21; Test type: Other; p = 0.0737, ANOVA
Statistical Analysis 8: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day21; Test type: Other; p = 0.2804, ANOVA

22. Primary Outcome: AUC0-8 for Paclitaxel
Description: as for outcome 18
Time Frame: Days -3 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours), 1 (0, 0.5, 1, 2, 4, 8, 24 hours), 8 (0, 0.5, 1, 2, 4, 8, 24 hours).
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: hr*microg/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
hr*microg/mL
  paclitaxel - AUC0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  paclitaxel - AUC0-8 - Day 1 | 4.05 (0.83) | 3.70 (0.89) | 5.82 (2.18)
  paclitaxel - AUC0-8 - Day 8: number analyzed (Participants) | 3 | 3 | 10
  paclitaxel - AUC0-8 - Day 8 | 3.70 (0.73) | 5.17 (3.08) | 5.69 (1.58)
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Paclitaxel, AUC0-8, Day 1; Test type: Other; p = 0.1449, ANOVA
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day 1; Test type: Other; p = 0.1338, ANOVA
Statistical Analysis 3: Comparison: Group 1 vs Group 3; Ibuprofen, AUC0-8, Day 8; Test type: Other; p = 0.0633, ANOVA
Statistical Analysis 4: Comparison: Group 2 vs Group 3; Ibuprofen, AUC0-8, Day 8; Test type: Other; p = 0.6939, ANOVA

23. Primary Outcome: Rac0-8 for DF1681Y
Description: PK parameters were calculated for cycle 1 only. Rac AUC0-8 is the Accumulation ratio calculated as the ratio of Day 8 to Day 1 AUC0-8.
Time Frame: Days 1 (0, 0.5, 1, 2, 4, 8, 24 hours), 8 (0, 0.5, 1, 2, 4, 8, 24 hours), and 21 (0, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours) of cycle 1
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ratio
  DF1681Y- Rac0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF1681Y- Rac0-8 - Day 1 | 0.97 (0.14) | 1.3 (0.53) | 1.21 (0.41)
  DF1681Y - Rac0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF1681Y - Rac0-8 - Day 8 | 0.63 (0.39) | 1.7 (0.88) | 1.01 (0.30)
  DF1681Y- Rac0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF1681Y- Rac0-8 - Day 21 | 0.82 (0.22) | 1.61 (0.63) | 1.02 (0.21)

24. Primary Outcome: Rac0-8 for DF2243Y
Description: as for outcome 23
Time Frame: as for outcome 23
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ratio
  DF2243Y- Rac0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2243Y- Rac0-8 - Day 1 | 1.02 (0.28) | 1.82 (1.06) | 1.18 (0.27)
  DF2243Y - Rac0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2243Y - Rac0-8 - Day 8 | 0.78 (0.64) | 1.3 (0.37) | 1.08 (0.23)
  DF2243Y- Rac0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2243Y- Rac0-8 - Day 21 | 1.15 (0.19) | 1.44 (0.11) | 1.16 (0.17)

25. Primary Outcome: Rac0-8 for DF2188Y
Description: as for outcome 23
Time Frame: as for outcome 23
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ratio
  DF2188Y- Rac0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  DF2188Y- Rac0-8 - Day 1 | 1.12 (0.34) | 1.61 (0.40) | 1.52 (0.51)
  DF2188Y - Rac0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  DF2188Y - Rac0-8 - Day 8 | 0.77 (0.54) | 1.32 (0.22) | 1.22 (0.27)
  DF2188Y- Rac0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  DF2188Y- Rac0-8 - Day 21 | 1.04 (0.09) | 1.35 (0.15) | 0.95 (0.15)

26. Primary Outcome: Rac0-8 for Ibuprofen
Description: as for outcome 23
Time Frame: as for outcome 23
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 12
ratio
  Ibuprofen - Rac0-8 - Day 1: number analyzed (Participants) | 4 | 3 | 11
  Ibuprofen - Rac0-8 - Day 1 | 1.09 (0.22) | 1.99 (1.38) | 1.18 (0.43)
  Ibuprofen - Rac0-8 - Day 8: number analyzed (Participants) | 4 | 3 | 10
  Ibuprofen - Rac0-8 - Day 8 | 0.65 (0.61) | 1.25 (0.28) | 1.23 (0.30)
  Ibuprofen - Rac0-8 - Day 21: number analyzed (Participants) | 3 | 3 | 8
  Ibuprofen - Rac0-8 - Day 21 | 1.18 (0.74) | 1.89 (0.86) | 1.24 (0.26)

27. Primary Outcome: Rac0-24 for Paclitaxel
Description: PK parameters were calculated for cycle 1 only. Rac AUC0-24 is the Accumulation ratio calculated as the ratio of Day 8 to Day 1 AUC0-24.
Time Frame: Day 8 (0, 0.5, 1, 2, 4, 8, 24 hours)
Population: PK Population: patients who received one dose of reparixin and had at least one valid, quantifiable PK parameter
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 3 | 3 | 10
ratio | 0.90 (0.110) | 1.59 (1.325) | 1.04 (0.121)

28. Secondary Outcome: Count of Patients With Complete Response (CR), Partial Response (PR), Stable Disease (SD), Disease Progression (PD) at Each Assessment Visit
Description: Complete Response/Remission(CR): Disappearance of all target lesions. Partial Response/Remission (PR): At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD.
  Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started.
  Progression of Disease (PD): At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At tumor assessments 1-11 and off-treatment visit
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
Participants
  Assessment 1 - CR | 1 | 0 | 0
  Assessment 1 - PR | 0 | 1 | 3
  Assessment 1 - SD | 0 | 0 | 9
  Assessment 1 - PD | 1 | 1 | 6
  Assessment 1.1 - CR | 0 | 0 | 0
  Assessment 1.1 - PR | 0 | 1 | 1
  Assessment 1.1 - SD | 0 | 0 | 0
  Assessment 1.1 - PD | 0 | 1 | 0
  Assessment 2 - CR | 1 | 0 | 0
  Assessment 2 - PR | 0 | 0 | 6
  Assessment 2 - SD | 0 | 0 | 2
  Assessment 2 - PD | 0 | 0 | 2
  Assessment 2.1 - CR | 0 | 0 | 0
  Assessment 2.1 - PR | 0 | 0 | 2
  Assessment 2.1 - SD | 0 | 0 | 0
  Assessment 2.1 - PD | 0 | 0 | 0
  Assessment 3 - CR | 1 | 0 | 0
  Assessment 3 - PR | 0 | 0 | 4
  Assessment 3 - SD | 0 | 0 | 0
  Assessment 3 - PD | 0 | 0 | 1
  Assessment 4 - CR | 1 | 0 | 1
  Assessment 4 - PR | 0 | 0 | 2
  Assessment 4 - SD | 0 | 0 | 0
  Assessment 4 - PD | 0 | 0 | 1
  Assessment 5 - CR | 1 | 0 | 1
  Assessment 5 - PR | 0 | 0 | 1
  Assessment 5 - SD | 0 | 0 | 0
  Assessment 5 - PD | 0 | 0 | 1
  Assessment 6 - CR | 1 | 0 | 1
  Assessment 6 - PR | 0 | 0 | 1
  Assessment 6 - SD | 0 | 0 | 0
  Assessment 6 - PD | 0 | 0 | 0
  Assessment 7 - CR | 1 | 0 | 0
  Assessment 7 - PR | 0 | 0 | 0
  Assessment 7 - SD | 0 | 0 | 0
  Assessment 7 - PD | 0 | 0 | 0
  Assessment 8 - CR | 1 | 0 | 0
  Assessment 8 - PR | 0 | 0 | 0
  Assessment 8 - SD | 0 | 0 | 0
  Assessment 8 - PD | 0 | 0 | 0
  Assessment 9 - CR | 1 | 0 | 0
  Assessment 9 - PR | 0 | 0 | 0
  Assessment 9 - SD | 0 | 0 | 0
  Assessment 9 - PD | 0 | 0 | 0
  Assessment 10 - CR | 1 | 0 | 0
  Assessment 10 - PR | 0 | 0 | 0
  Assessment 10 - SD | 0 | 0 | 0
  Assessment 10 - PD | 0 | 0 | 0
  Assessment 11 - CR | 1 | 0 | 0
  Assessment 11 - PR | 0 | 0 | 0
  Assessment 11 - SD | 0 | 0 | 0
  Assessment 11 - PD | 0 | 0 | 0
  Off-treatment visit - CR | 1 | 0 | 1
  Off-treatment visit - PR | 0 | 0 | 1
  Off-treatment visit - SD | 0 | 0 | 1
  Off-treatment visit - PD | 1 | 1 | 8

29. Secondary Outcome: Best Overall Response (BOR)
Description: The best overall response (BOR) was defined as the number of patients reaching complete remission (CR), partial remission (PR) or stable disease (SD) according to RECIST criteria version 1.1
Time Frame: After 24 weeks
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
Participants
  CR | 1 | 0 | 1
  PR | 0 | 0 | 5
  SD | 0 | 1 | 7
  PD | 2 | 2 | 7

30. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The clinical benefit rate (CBR) was defined as the percentage of patients reaching CR, PR or SD according to RECIST criteria version 1.1
Time Frame: After 24 weeks
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Number; unit: Percentage of patients
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
Percentage of patients | 25.0 | 33.3 | 56.5

31. Secondary Outcome: 6-month Progression-free Survival Rate
Description: The 6-month progression-free survival rate (%) was defined as the percentage of patients with no mortality and at least 24-week duration of CR, PR or SD according to RECIST criteria version 1.1
Time Frame: After 24 weeks
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Number; unit: Percentage of patients
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
Percentage of patients | 25.0 | 0.0 | 17.4

32. Secondary Outcome: Median Time to Tumor Progression in Days (TTP)
Description: The median time to tumor progression in days (TTP) was defined as the time from the date of the first administration of study drug to the date of the first documentation of progressive disease
Time Frame: After 24 weeks
Population: Safety Population: all enrolled patients who took at least one dose of study drug, reparixin.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 4 | 3 | 23
days | 58 [44 to NA] — the sample size of group 1 does not allow the calculation of the upper bound of the confidence interval | 67 [58 to NA] — the sample size of group 2 does not allow the calculation of the upper bound of the confidence interval | 170 [65 to 229]

ADVERSE EVENTS:
Time Frame: Throughout the study from run-in to off-treatment visit, up to 24 months.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 4/23
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=4) | Group 2 (N=3) | Group 3 (N=23)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=4) | Group 2 (N=3) | Group 3 (N=23)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (9) | 10 (12)
Nausea (Gastrointestinal disorders) | 3 (5) | 3 (13) | 12 (16)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 8 (13)
Vomiting (Gastrointestinal disorders) | 3 (7) | 2 (4) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No